CLINICAL TRIAL: NCT04004455
Title: Exploring Pain, Body Composition and Physical Activity in Childhood Cancer: a Case Control Study
Brief Title: Pain, Body Composition and Physical Activity in Childhood Cancer.
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Emma Rheel, PhD student, Vrije Universiteit Brussel
Other Study IDs: CASECONTROL_RE_2019-2020
Record Dates: First submitted 2019-06-19; First posted 2019-07-02 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Childhood Cancer
Keywords: children; cancer; pressure pain threshold; energy-balance related behavior; pain catastrophizing; body composition
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Childhood cancer: Children with an established cancer diagnosis (any type) between 8-18 years old that are currently being treated for cancer (not necessarily hospitalized) in the University Hospital Brussels or Ghent.
- Healthy controls: Healthy children between 8-12 years old, selected based on age and sex.

SUMMARY:
Comparing baseline assessments of children with cancer and their parents with baseline assessments of healthy children and their parents in a case-control study will allow the investigators to make the comparison in terms of pressure hyperalgesia, pain catastrophizing, energy-balance related behavior, attention control and attention bias between healthy children and cancer patients. This also enables the investigators to compare parents of healthy children with parents of cancer patients in the field of catastrophizing about the pain of their child and responses to child's pain experiences. Correlations can also be calculated between, for example, pain pressure thresholds and energy-balance related behavior.

DETAILED DESCRIPTION:
Participant recruitment

Cancer patients will be recruited by the oncology department of the children's hospital of the University Hospital Brussels and Ghent. All children with cancer between 8-18y and their parents will be informed about the study and receive a consent form. The recruitment procedure will start in July 2019 and pursue until the calculated sample size is reached. Healthy controls will be recruited from several schools in the neighborhood and from family and acquaintances of the hospital personnel and researchers. In order to be able to compare their outcomes with the intervention group, they will be selected based on age and sex. Cancer patients with a portal catheter will also be included in a concurrent pilot randomized controlled trial, including the same baseline assessments. In this pilot randomized controlled trial, children will be distracted by a humanoid robot during painful medical procedures. Given the observation that children up to 12 years of age are more likely than children over 12 years to believe that a robot possesses human characteristics, only the children between the ages of 8 and 12 years also participate in this randomized controlled trial. The lower age limit is chosen because child self-report questionnaires have been validated from that age. Self-reports in children also require a variety of cognitive skills, which develop gradually and are only acquired at the age of 7 or 8 in most children. Children and their parents can only be included in the study if they meet the inclusion criteria and after written informed consent from the (co-participating) parent/guardian and child is obtained. All parents/guardians and children will receive verbal and written information on all aspects of the study prior to consent for participation.

Sample size calculation was performed with G*Power 3.1.9.2 (Franz Faul, Kiel, Germany). The a priori sample size calculation for this study was based on the sample size calculation of a previous study on pain hypersensitivity in juvenile idiopathic arthritis compared with healthy children. Targeting a study power of 80% with an α error probability of 0.05 and allocation ratio (N1/N2) defined as 1, the calculation revealed sample sizes of 26 participants for the cancer group and 26 participants for the healthy controls (total sample size n=52). Accounting for a 10% dropout and keeping in mind that every sample size calculation has its limitations, the investigators propose studying at least 30 participants per group. Hence, the total number of participants to be included will be equal to 60. Because of the low number of new cases of childhood cancer (<15 years of age) per year in Belgium, the monocentric nature of this trial and the limited time for data collection (1 year 9 months) the calculated sample size remains as a target.

Risk management: In case of slow patient recruitment or a dropout rate that exceeds 10%, the age range of the participants will be extended (1) and French speaking children and their parents will no longer be excluded (2).

Assessments

Using an online questionnaire battery (↑ study feasibility), a number of measures will be assessed in the participating children and their parent(s). Online questionnaires will set up with Lime Survey.

Demographics and medical data:

Demographics (e.g. age, sex, ethnicity, socioeconomic status) and medical information will be collected from the patient's clinical charts and will be further supplemented by child and parent report.

Anthropometrics:

Basic anthropometrics (body height, body weight, waist circumference) will be gathered from each participating child. In addition, the body composition (i.e., body mass index, fat mass, fat free mass, muscle mass, intra- and extra cellular water, etcetera) will be determined by 1 body composition analyzer (and an additioinial one in the healthy control group).

Pressure hyperalgesia: pressure pain threshold (PPT) - CHILD:

Pressure hyperalgesia of all participating children will be assessed by evaluating pressure pain thresholds (PPTs) at the dominant tibialis anterior and trapezius muscle by means of a digital pressure algometer (FPX 50, Wagner Instruments, Greenwich, CT, USA). To familiarize the subject with PPT measurements, one familiarization session will be done at the dominant upper leg. This technique to evaluate PPTs is a well-known and well validated method in the exploration of pathophysiological mechanisms involved in pain. High reliability levels of this technique are apparent from various studies. Also, pressure algometry has proven to have an excellent intra-rater agreement, a satisfactory inter-rater agreement and is well tolerated even by very young children.

Pain catastrophizing Scale for Children (PCS-C) - CHILD:

Children's catastrophic thinking about pain will be assessed with the Dutch version of the Pain Catastrophizing Scale for Children (PCS-C). The PCS-C consists of 13 items describing thoughts and feelings which the child may experience when they are in pain, in independent but strongly related dimensions of rumination, magnification and helplessness. Children are asked to rate how frequently they experience these thoughts and feelings on a 5-point Likert scale (0 = 'not at all', 4 = 'extremely'). The PCS-C results in a total score (ranging from 0 to 52). The PCS-C has been shown to be a reliable and valid tool for children of 9 to 15 years old and a strong internal consistency for pain catastrophizing (α=.90) is already demonstrated in the pediatric population.

Attentional Control Scale for Children (ACS-C) - CHILD:

Attention control will be assessed using the Attentional Control Scale for Children (ACS-C), which is a 20 item self-rating scale that assesses abilities to focus and shift attention. Ten statements assess the focusing component of attention (''When I concentrate myself, I do not notice what is happening in the room around me'') and the other ten statements assess the shifting of attentional resources (''When I am doing something, I can easily stop and switch to some other task''). A higher score on this scale indicates a better capacity of attentional control. Several studies report good internal consistency of the ACS-C.

Attention Bias Assessment (dot-probe task) - CHILD:

All participating children will be asked to complete a dot-probe task, which is a well-investigated reaction time task designed to measure selective attention to threat. In this dot-probe task, a threatening (i.e., pain) and neutral stimulus are presented simultaneously (i.e., a painful child face paired with a neutral child face) at two different spatial locations on a screen for a short time. Because both stimuli are in different spatial locations, they compete for attention. After the appearance of these stimuli, a dot probe emerges at the location of the threatening/pain stimulus (congruent presentation) or at the location of the neutral stimulus (incongruent presentation). The assignment of attention is measured by the time needed to respond to the dot probe. It is reasoned that responding to the probe will be faster when the child's attention is already allocated to location where the probe appears. Most probe detection studies found indeed that anxious individuals respond faster to congruent trials than to incongruent trials (congruency effect). This task is implicit, does not require instruction, and subjects need no or minimal training to perform the test successfully.

Energy balance-related behavior (ENERGY Cross Sectional Survey (CSS) child) - CHILD:

A selection of questions regarding physical activity and sedentary behavior of the ENERGY Cross-Sectional Survey (ENERGY CSS child) used in the ENERGY-project will be assessed by the participating children. This ENERGY-child questionnaire was developed in order to assess energy balance-related behaviors of the child as well as personal, family and school-environmental determinants related to these behaviors. The questionnaire has been shown to have good test-retest reliability and moderate to good construct validity for the large majority of items.

Pain Catastrophizing Scale for Parents (PCS-P) - PARENT:

Parent's catastrophic thinking about their child's pain will be assessed with the Dutch version of the Pain Catastrophizing Scale for Parents (PCS-P). The PCS-P consists of 13 items describing different thoughts and feelings that parents may experience in relation to their child's pain, in independent but strongly related dimensions of rumination, magnification and helplessness. Parents are asked to rate how frequently they experience these thoughts and feelings on a 5-point Likert scale (0 = 'not at all', 4 = 'extremely'). The developers reported strong internal consistency (α=.93) and validity as demonstrated by associations with parent distress and child disability.

Inventory of parent/caregiver responses to the children's pain experience (IRPEDNA) - PARENT:

To measure the responses of the parent to their child's pain episodes at T0, a shortened of the inventory of parent/caregiver responses to the children's pain experience (IRPEDNA) will be used. The scale is a self-administered questionnaire with three subscales: (1) solicitousness, (2) discouragement, and (3) promotion of well-behaviors and coping. The shortened version of 10 items only includes solicitousness and promotion of well-behaviors. All items reflect actions and behaviors that the parents may enact after seeing the children's pain behaviors. A good internal consistency of the 3 subscales has been demonstrated (coefficient alphas of 0.87, 0.83 and 0.87 respectively) and the subscales also show good criterion-related validity.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Willing to participate and comply with pre-determined interventions
* 8-18y (children)
* Child and parent(s)/guardian cohabited for the past 5 years or, in case of divided custody, for at least half of the child's lifetime

Cancer patients

* Established cancer diagnosis (any type)
* First cancer diagnosis
* Currently being treated for cancer (not necessarily hospitalized) in the University Hospital Brussels or Ghent

Exclusion Criteria:

* Developmental disabilities (e.g.: autism spectrum disorder, Attention Deficit (Hyperactivity) Disorder)
* Psychiatric disorders (e.g.: anxiety disorder, personality disorder)
* Significant vision or hearing impairment
* Chronic pain diagnosis (e.g.: fibromyalgia, migraine, chronic abdominal pain, etc.)
* Not able to read and speak fluent Dutch (parent and child)
* Already having undergone any kind of self-regulation and/or behavioral therapy for pain (i.e. relaxation, hypnosis, biofeedback, pain neuroscience education, cognitive behavioral therapy, etc.)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cancer patients will be recruited by the oncology department of the children's hospital of the University Hospital Brussels and Ghent. All eligibel children between 8-18y and their parents will be informed about the study and receive a consent form. Healthy controls will be recruited from several schools in the neighborhood and from family and acquaintances of the hospital personnel and researchers. In order to be able to compare their outcomes with the intervention group, they will be selected based on age and sex.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Pressure hyperalgesia (child) | 1 day
  Pain response to stimuli that are normally not painful, induced by the lowering of the nociceptor threshold level and assessed by evaluating pressure pain thresholds (PPTs) at the dominant tibialis anterior and trapezius muscle by means of a digital pressure algometer (FPX 50, Wagner Instruments, Greenwich, CT, USA). Per test site, 3 measurements are performed with 30 seconds between each measurement. The measurements take place alternately between the two test sites, the first test site being randomly determined by an independent blinded researcher. The pressure pain threshold in kgf per muscle (test site) is determined by the mean of the 2nd and 3rd measurement.

SECONDARY OUTCOMES:
Energy-balance related behavior (child) | 1 day
  Physical activity and screen behavior. A selection of questions regarding physical activity (E1-E12) and sedentary behavior (F1-F2) of the ENERGY Cross-Sectional Survey (ENERGY CSS child) will be assessed by the participating children.
Waist circumference (child) | 1 day
  Waist circumference of the child in centimeters, measured at umbilical level and at 4 centimeters above the umbilicus.
Body length (child) | 1 day
  Body length of the child in centimeters.
Body weight (child) | 1 day
  Body weight of the child in kilograms, determined with the TANITA MC-780SMA (from Tanita Corporation).
Body weight (only healthy controls) (child) | 1 day
  Body weight in kilograms of the children in the healthy control group will also be determined with the OMRON VIVA (OMRON VIVA HBF-222T-EBK from OMRON Healthcare Co).
Fat percentage (child) | 1 day
  Body fat percentage of the child, determined with the TANITA MC-780SMA (from Tanita Corporation).
Fat percentage (only healthy controls) (child) | 1 day
  Body fat percentage of the children in the healthy control group will also be determined with the OMRON VIVA (OMRON VIVA HBF-222T-EBK from OMRON Healthcare Co).
Fat mass (child) | 1 day
  Fat mass of the child in kilograms, determined with the TANITA MC-780SMA (from Tanita Corporation).
Fat free mass (child) | 1 day
  Fat free mass of the child in kilograms, determined with the TANITA MC-780SMA (from Tanita Corporation).
Muscle mass (child) | 1 day
  Muscle mass of the child in kilograms, determined with the TANITA MC-780SMA (from Tanita Corporation).
Muscle mass percentage (only healthy controls) (child) | 1 day
  Muscle mass percentage of the children in the healthy control group will be determined with the OMRON VIVA (OMRON VIVA HBF-222T-EBK from OMRON Healthcare Co).
Total body water (child) | 1 day
  Total body water of the child in kilograms, determined with the TANITA MC-780SMA (from Tanita Corporation).
Total body water percentage (child) | 1 day
  Total body water percentage of the child, determined with the TANITA MC-780SMA (from Tanita Corporation).
Intracellular water (child) | 1 day
  Intracellular water (ICW) of the child in kilograms, determined with the TANITA MC-780SMA (from Tanita Corporation).
Extracellular water (child) | 1 day
  Extracellular water (ECW) of the child in kilograms, determined with the TANITA MC-780SMA (from Tanita Corporation).
Body mass index (child) | 1 day
  Body mass index of the child in kilograms/m^2, determined with the TANITA MC-780SMA (from Tanita Corporation).
Body mass index (only healthy controls) (child) | 1 day
  Body mass index of the child in kilograms/m^2, determined with the OMRON VIVA (OMRON VIVA HBF-222T-EBK from OMRON Healthcare Co).
Visceral fat rating (child) | 1 day
  Visceral fat rating of the child on a scale from 1 to 59, determined with the TANITA MC-780SMA (from Tanita Corporation).
Visceral fat rating (only healthy controls) (child) | 1 day
  Visceral fat rating i(n 30 levels) of the children in the healthy control group will also be determined with the OMRON VIVA (OMRON VIVA HBF-222T-EBK from OMRON Healthcare Co).
Basal metabolic rate (child) | 1 day
  Basal metabolic rate of the child in kcal, determined with the TANITA MC-780SMA (from Tanita Corporation).
Basal metabolic rate (only healthy controls) (child) | 1 day
  Basal metabolic rate of the children in the healthy control group in kcal, determined with the OMRON VIVA (OMRON VIVA HBF-222T-EBK from OMRON Healthcare Co).
Attention control child (child) | 1 day
  Attention control is defined as an individual's capacity to choose what they pay attention to and what they ignore. Attention control will be assessed using the Attentional Control Scale for Children (ACS-C), which is a 20 item self-rating scale that assesses abilities to focus and shift attention. Ten statements assess the focusing component of attention (''When I concentrate myself, I do not notice what is happening in the room around me'') and the other ten statements assess the shifting of attentional resources (''When I am doing something, I can easily stop and switch to some other task''). The child rates each question on a 4 point Likert scale (1 = almost never to 4 = always).
Attention bias (child) | 1 day
  Attention bias is defined as a selective attention to threat. All participating children will be asked to complete a dot-probe task, which is a well-investigated reaction time task designed to measure selective attention to threat. In this dot-probe task, a threatening (i.e., pain) and neutral stimulus are presented simultaneously (i.e., a painful child face paired with a neutral child face) at two different spatial locations on a screen for a short time. After the appearance of these stimuli, a dot probe emerges at the location of the threatening/pain stimulus (congruent presentation) or at the location of the neutral stimulus (incongruent presentation). The attentional bias is the response time to incongruent trials minus the response time to congruent trials: a positive index indicates more attention to pain; a negative index indicates attentional avoidance.
Responses to child's pain experience (parent) | 1 day
  To measure the responses of the parent to their child's pain episodes, a shortened version of the inventory of parent/caregiver responses to the children's pain experience (IRPEDNA) will be used. The original scale is a self-administered questionnaire with three subscales: (1) solicitousness, (2) discouragement, and (3) promotion of well-behaviors and coping. The shortened version will only include subscale 1 and 3. All 10 items of the shortened version reflect actions and behaviors that the parents may enact after seeing the children's pain behaviors. Participating parents rate each item using a five-point response scale (1, never; 2, hardly ever; 3, sometimes; 4, often; 5, always), with final scores ranging from 10 to 50.

OTHER OUTCOMES:
Pain catastrophizing (child) | 1 day
  Thoughts and feelings which the child may experience when they are in pain. Children's catastrophic thinking about pain will be assessed with the Dutch version of the Pain Catastrophizing Scale for Children (PCS-C). The scale consists of 13 items describing different thoughts and feelings that children may experience when they are in pain. Children are asked to rate how frequently they experience these thoughts and feelings on a 5-point Likert scale (0 = 'not at all', 4 = 'extremely'). The PCS-C results in a total score (ranging from 0 to 52), and three subscale scores for rumination, magnification and helplessness.
Pain catastrophizing (parent) | 1 day
  Thoughts and feelings that parents may experience in relation to their child's pain. Parent's catastrophic thinking about their child's pain will be assessed with the Dutch version of the Pain Catastrophizing Scale for Parents (PCS-P). Similar to the PCS-C, the PCS-P consists of 13 items describing different thoughts and feelings that parents may experience in relation to their child's pain. Parents are asked to rate how frequently they experience these thoughts and feelings on a 5-point Likert scale (0 = 'not at all', 4 = 'extremely'). The PCS-P results in a total score (ranging from 0 to 52), and three subscale scores for rumination, magnification and helplessness.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brussels, Jette, Brussels Capital, Belgium